CLINICAL TRIAL: NCT06008067
Title: The Prognostic Role of Tricuspid Annular Plane Systolic Excursion in Critically Ill Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: TAPSESEPTIC
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Septic Shock
Keywords: Critical Care; Septic Shock; Echocardiography; RV dysfunction
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Patients who survived after day 28.
  Interventions: Radiation: tricuspid annular plane systolic excursion (TAPSE)
- Non-survivors: Patients who died at or before day 28.
  Interventions: Radiation: tricuspid annular plane systolic excursion (TAPSE)

INTERVENTIONS:
Radiation: tricuspid annular plane systolic excursion (TAPSE) — Echocardiography

SUMMARY:
The aim of this study is to evaluate the possible prognostic performance of RV dysfunction, as assessed by TAPSE, in non-cardiac patients with septic shock.

DETAILED DESCRIPTION:
The objective is to investigate the prognostic performance of right ventricular dysfunction, as assessed by tricuspid annular plane systolic excursion (TAPSE), in non-cardiac patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 - 64 years old) with septic shock after admission according to 2016 consensus definition (Sepsis-3).

Exclusion Criteria:

* Pregnant females
* Trauma
* Documented coronary heart disease
* History of myocardial infarction
* Myocarditis
* Thrombo-embolic pulmonary disease
* Valvular heart disease
* Corpulmonale
* Arrhythmia
* Known left ventricular ejection fraction < 40%
* Poor echocardiographic window

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Adult patients (18 - 64 years old) with septic shock after admission according to 2016 consensus definition (Sepsis-3).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
28-day mortality | Day 28
  Mortality rate after at day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Habib, MD, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine, Alexandria University Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habib T, Ahmed I, Abayazeed R, Montasser M. The prognostic role of tricuspid annular plane systolic excursion in critically ill patients with septic shock. J Anesth Analg Crit Care. 2025 Apr 30;5(1):24. doi: 10.1186/s44158-025-00227-0. PMID 40307938